CLINICAL TRIAL: NCT02728310
Title: Local Continuous Wound Infusion and Local Infusion of Anaesthetics in the Management of Post-operative Pain and Rehabilitation After Total Hip Arthroplasty: a Double-blind Randomized Controlled Clinical Trial
Brief Title: Local Continuous Wound Infusion of Anesthetics in the Management of Post-operative Pain After Total Hip Arthroplasty.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, Anesthesist, San Salvatore Hospital of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0080580/12
Record Dates: First submitted 2016-03-15; First posted 2016-04-05 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Levobupivacaine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levobupivacaine infusion (Active Comparator): 1500 mg of Levobupivacaine by an infusion rate of 10 ml/h for the first 30 h and 5 ml/h for the second 30 h (LCWI) were injected.
  Interventions: Drug: Levobupivacaine
- Saline infusion (Placebo Comparator): 300 ml of Saline (for Levobupivacaine as placebo) by an infusion rate of 10 ml/h for the first 30 h and 5 ml/h for the second 30 h (LCWI) were injected.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Levobupivacaine — An infusion rate of 10 ml/h of 1500 mg of 0.5 % of levobupivacaine for the first 30 h and 5 ml/h for the second 30 h (LCWI) were injected into the surgical wound.
  Other Names: Chiracaine
  Arms: Levobupivacaine infusion
Drug: Saline — An infusion rate of 10 ml/h of 300 ml of saline solution for the first 30 h and 5 ml/h for the second 30 h (LCWI) were injected into the surgical wound.
  Other Names: Saline solution
  Arms: Saline infusion

SUMMARY:
The combination of subarachnoid anaesthesia (SAB) and continuous local wound infiltration (LCWI) with a consistent amount of local anaesthetics could prevent central sensitization through an additive or synergistic effect because it can maintain continuous inhibition of nociceptive afferents

DETAILED DESCRIPTION:
Wound infiltration with local anesthetics is an analgesic technique that has been adopted for post-operative analgesia following a range of surgical orthopaedic procedures. Pain management by infusion of local aesthetic into wounds was found to improve pain, reduced opioid use and side effects, increase patient satisfaction, and shorten the hospital stay when compared to placebo or no treatment, but actually it was not definitively proven that wound infiltration provides additional analgesic or outcome benefit in the setting of a comprehensive multimodal analgesic approach. The hypothesis of this study is that a consistent amount of Levobupivacaine 0.5% for LCWI and LIA could provide a more extended postoperative analgesia for post-operative incident and rest pain with a better post-operative recovery and rehabilitation following THA, in the first 72 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years of age
* American Society of Anaesthesiologists (ASA) physical status I-III
* total hip arthroplasty.

Exclusion Criteria:

* pregnancy
* body mass index (BMI) >35
* allergy to local anaesthetics
* skeletal and/or muscle abnormalities of the spine
* primary and/or secondary neurological diseases
* psychiatric diseases
* history of chronic pain and/or neuropathic disorders
* history of drug abuse
* state of sepsis
* infection and/or tumours within the skin on the back
* primary or secondary coagulopathies
* primary or secondary heart, liver and renal failure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Incident and rest pain (using VAS score) at 72 hours after surgery | 72 hours
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Consumption of painkillers (in mg) at 72 hours after surgery | 72 hours
  The equianalgesic dose (in mg) of morphine
Side effects (PONV) at 72 hours after surgery | 72 hours
  Time to have post-operative nausea and vomiting (in minutes)
Toxicity of local anaesthetics (epilepsy) at 72 hours after surgery | 72 hours
  Presence or not of epilepsy
Wound healing at 72 hours | 72 hours
  Number of infections of surgical wound.
Improvement of rehabilitation at 72 hours | 72 hours
  Our total hip arthroplasy rehabilitation protocol is focused on the following manoeuvres: contraction of the gluteal and quadricipital muscles, passive and active mobilization of the hip joint, passive and active mobilization of the knee and walking with crutches and a walker.the improvement of rehabilitation manoeuvres has been evaluated in a four-step scale: 0-no improvement; 1- slight improvement, 2- good improvement; 3- great improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Pierfrancesco Fusco, MD, Principal Investigator — Anesthesia and Intensive care Unit, San Salvatore Academic Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konopka JF, Hansen VJ, Rubash HE, Freiberg AA. Risk assessment tools used to predict outcomes of total hip and total knee arthroplasty. Orthop Clin North Am. 2015 Jul;46(3):351-62, ix-x. doi: 10.1016/j.ocl.2015.02.004. Epub 2015 Mar 24. PMID 26043049
- [Result] Di Puccio F, Mattei L. Biotribology of artificial hip joints. World J Orthop. 2015 Jan 18;6(1):77-94. doi: 10.5312/wjo.v6.i1.77. eCollection 2015 Jan 18. PMID 25621213